CLINICAL TRIAL: NCT00861380
Title: Evaluation of Effectiveness of GSK Biologicals' Pneumococcal Conjugate Vaccine 1024850A Against Invasive Disease
Acronym: FinIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 111442; 2008-005149-48 (EudraCT Number)
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Infections, Streptococcal; Streptococcus Pneumoniae
Keywords: Pneumococcal conjugate vaccine; Invasive disease; Respiratory tract infections; Haemophilus influenzae; Streptococcus pneumoniae; Acute otitis media; Pneumonia
MeSH Terms: conditions — Streptococcal Infections; Respiratory Tract Infections; Haemophilus Infections; Otitis Media; Pneumonia | interventions — Hepatitis B Vaccines; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- 10Pn3+1-6W- 6M/043 Group (Experimental): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) study, aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule). The vaccine was administered intramuscularly in the thigh.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A
- 10Pn2+1-6W-6M/043 Group (Experimental): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) study, aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). The vaccine was administered intramuscularly in the thigh.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A
- Ctrl-6W-6M/043 Group (Active Comparator): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) study, aged 6 weeks to 6 months at enrolment. Subjects received the Engerix B vaccine (called also HBV vaccine) according to either a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule), or according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). The vaccine was administered intramuscularly in the thigh.
  Interventions: Biological: GSK Biologicals' Engerix TM vaccine (Hepatitis B vaccine)
- 10Pn7-11M/043 Group (Experimental): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) study, aged 7 to 11 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (11-17M Schedule). The vaccine was administered intramuscularly in the thigh or in the deltoid region of upper arm, provided the muscle size was adequate.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A
- Ctrl7-11M/043 Group (Active Comparator): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) study, aged 7 to 11 months at enrolment. Subjects received the Engerix B (called also HBV) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (11-17M Schedule). The vaccine was administered intramuscularly in the thigh or in the deltoid region of upper arm, provided the muscle size was adequate.
  Interventions: Biological: GSK Biologicals' Engerix TM vaccine (Hepatitis B vaccine)
- 10Pn12-18M/043 Group (Experimental): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) study, aged 12 to 18 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). The vaccine was administered intramuscularly in the thigh or in the deltoid region of upper arm, provided the muscle size was adequate.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A
- Ctrl12-18M/043 Group (Active Comparator): Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) study, aged 12 to 18 months at enrolment. Subjects received the Havrix (called also HAV) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). The vaccine was administered intramuscularly in the thigh or in the deltoid region of upper arm, provided the muscle size was adequate.
  Interventions: Biological: GSK Biologicals' Havrix TM vaccine (Hepatitis A vaccine)

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine GSK1024850A — 2, 3 or 4 Intramuscular injections, depending on the age at the time of first vaccination
  Arms: 10Pn12-18M/043 Group; 10Pn2+1-6W-6M/043 Group; 10Pn3+1-6W- 6M/043 Group; 10Pn7-11M/043 Group
Biological: GSK Biologicals' Engerix TM vaccine (Hepatitis B vaccine) — 3 or 4 Intramuscular injections, depending on the age at the time of first vaccination.
  Control 3+1 and Control 2+1 groups, only for children < 12 months of age at the time of first study vaccination.
  Arms: Ctrl-6W-6M/043 Group; Ctrl7-11M/043 Group
Biological: GSK Biologicals' Havrix TM vaccine (Hepatitis A vaccine) — 2 Intramuscular injections. Control 3+1 and Control 2+1 groups, only for children >= 12 months of age at the time of first study vaccination.
  Arms: Ctrl12-18M/043 Group

SUMMARY:
The aim of this study is to assess the effectiveness of GSK Biologicals' pneumococcal conjugate vaccine (GSK1024850A), administered according to different vaccination schedules, against invasive disease caused by S. pneumoniae or H. influenzae as well as vaccine impact on the occurrence of hospital-diagnosed pneumonia cases, tympanostomy tube placement and outpatient antimicrobial prescriptions.

This study will also explore vaccine impact on occurrence of respiratory tract infections (RTIs), including acute otitis media (AOM) in a subset of children in Turku area.

DETAILED DESCRIPTION:
The protocol posting has been updated with regards to the enrolment of subjects and outcome measures following Protocol amendment 2, 22 August 2011.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between, and including, 6 weeks to 18 months of age at the time of the first vaccination.
* Written informed consent obtained from parent(s) or from the guardian(s) of the subject.

Exclusion Criteria:

* Previous vaccination with any registered, non-registered or investigational pneumococcal vaccine other than the study vaccine, or planned use during the study period. If a child belongs to a high risk group for pneumococcal infections for which a licensed pneumococcal conjugate vaccine is made locally available, the subject can not be enrolled in the study and should be referred to the specific immunization program.
* Previous vaccination against Hepatitis B virus with any registered, non-registered or investigational vaccine, or planned use of such a vaccine other than the study vaccine during the study period.
* Previous vaccination against Hepatitis A virus with any registered, non-registered or investigational vaccine, or planned use of such a vaccine other than the study vaccine during the study period.
* Known severe hypersensitivity to any component of the study vaccines, including neomycin.
* Any medical condition that would contraindicate the initiation of routine immunization outside a clinical trial context.

Ages: 6 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41188 (Actual)
Dates: Start 2009-05-04 (Actual); Primary Completion 2012-01-31 (Actual); Study Completion 2013-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=261

REFERENCES:
- [Background] Palmu AA, Jokinen J, Borys D, Nieminen H, Ruokokoski E, Siira L, Puumalainen T, Lommel P, Hezareh M, Moreira M, Schuerman L, Kilpi TM. Effectiveness of the ten-valent pneumococcal Haemophilus influenzae protein D conjugate vaccine (PHiD-CV10) against invasive pneumococcal disease: a cluster randomised trial. Lancet. 2013 Jan 19;381(9862):214-22. doi: 10.1016/S0140-6736(12)61854-6. Epub 2012 Nov 16. PMID 23158882
- [Background] Palmu AA, Jokinen J, Nieminen H, Rinta-Kokko H, Ruokokoski E, Puumalainen T, Borys D, Lommel P, Traskine M, Moreira M, Schuerman L, Kilpi TM. Effect of pneumococcal Haemophilus influenzae protein D conjugate vaccine (PHiD-CV10) on outpatient antimicrobial purchases: a double-blind, cluster randomised phase 3-4 trial. Lancet Infect Dis. 2014 Mar;14(3):205-12. doi: 10.1016/S1473-3099(13)70338-4. Epub 2013 Nov 26. PMID 24287186
- [Background] Palmu AA, Jokinen J, Nieminen H, Syrjanen R, Ruokokoski E, Puumalainen T, Moreira M, Schuerman L, Borys D, Kilpi TM. Vaccine effectiveness of the pneumococcal Haemophilus influenzae protein D conjugate vaccine (PHiD-CV10) against clinically suspected invasive pneumococcal disease: a cluster-randomised trial. Lancet Respir Med. 2014 Sep;2(9):717-27. doi: 10.1016/S2213-2600(14)70139-0. Epub 2014 Aug 7. PMID 25127244
- [Background] Palmu AA, Jokinen J, Nieminen H, Rinta-Kokko H, Ruokokoski E, Puumalainen T, Traskine M, Moreira M, Borys D, Schuerman L, Kilpi TM. Effectiveness of the Ten-valent Pneumococcal Conjugate Vaccine Against Tympanostomy Tube Placements in a Cluster-randomized Trial. Pediatr Infect Dis J. 2015 Nov;34(11):1230-5. doi: 10.1097/INF.0000000000000857. PMID 26284652
- [Background] Palmu AA, Jokinen J, Nieminen H, Rinta-Kokko H, Ruokokoski E, Puumalainen T, Moreira M, Schuerman L, Borys D, Kilpi TM. Vaccine-preventable disease incidence of pneumococcal conjugate vaccine in the Finnish invasive pneumococcal disease vaccine trial. Vaccine. 2018 Mar 27;36(14):1816-1822. doi: 10.1016/j.vaccine.2018.02.088. PMID 29503110
- [Background] Nieminen H, Rinta-Kokko H, Jokinen J, Puumalainen T, Moreira M, Borys D, Schuerman L, Palmu AA. Effectiveness of the 10-valent pneumococcal conjugate vaccine among girls, boys, preterm and low-birth-weight infants - Results from a randomized, double-blind vaccine trial. Vaccine. 2019 Jun 19;37(28):3715-3721. doi: 10.1016/j.vaccine.2019.05.033. Epub 2019 May 20. PMID 31122856
- [Background] Kilpi TM, Jokinen J, Puumalainen T, Nieminen H, Ruokokoski E, Rinta-Kokko H, Traskine M, Lommel P, Moreira M, Ruiz-Guinazu J, Borys D, Schuerman L, Palmu AA. Effectiveness of pneumococcal Haemophilus influenzae protein D conjugate vaccine against pneumonia in children: A cluster-randomised trial. Vaccine. 2018 Sep 18;36(39):5891-5901. doi: 10.1016/j.vaccine.2018.08.020. Epub 2018 Aug 23. PMID 30145098
- [Derived] Rinta-Kokko H, Palmu AA, Ruokokoski E, Nieminen H, Moreira M, Schuerman L, Borys D, Jokinen J. Evaluation of the indirect impact of the 10-valent pneumococcal Haemophilus influenzae protein D conjugate vaccine in a cluster-randomised trial. PLoS One. 2022 Jan 5;17(1):e0261750. doi: 10.1371/journal.pone.0261750. eCollection 2022. PMID 34986178
- [Derived] Vesikari T, Forsten A, Seppa I, Kaijalainen T, Puumalainen T, Soininen A, Traskine M, Lommel P, Schoonbroodt S, Hezareh M, Moreira M, Borys D, Schuerman L. Effectiveness of the 10-Valent Pneumococcal Nontypeable Haemophilus influenzae Protein D-Conjugated Vaccine (PHiD-CV) Against Carriage and Acute Otitis Media-A Double-Blind Randomized Clinical Trial in Finland. J Pediatric Infect Dis Soc. 2016 Sep;5(3):237-248. doi: 10.1093/jpids/piw010. Epub 2016 Apr 28. PMID 27125273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study also served as basis for conducting a long-term evaluation of the impact of vaccination with GSK Biologicals' 10Pn-PD-DiT vaccine. Subjects of the 10PN-PD-DIT-053 (112595) study (NCT00839254-EUDRACT:2008-006551-51) contributed to the objectives of this study.
Pre-assignment Details: 41188 subjects were enrolled in the study, 7 subjects didn't receive any vaccination, 41181 subjects started the study. Total population assessed for combined analyses performed on both studies included 45977 subjects, see details in groups description.
Groups:
- 10Pn3+1-6W-6M/043 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) study, aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule). The vaccine was administered intramuscularly in the thigh.
Period: Overall Study
Arm/Group | 10Pn3+1-6W-6M/043 Group | 10Pn2+1-6W-6M/043 Group | Ctrl-6W-6M/043 Group | 10Pn7-11M/043 Group | Ctrl7-11M/043 Group | 10Pn12-18M/043 Group | Ctrl12-18M/043 Group
Started | 8427 | 9112 | 8872 | 3689 | 1812 | 6249 | 3020
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8427 | 9112 | 8872 | 3689 | 1812 | 6249 | 3020
Not completed — Withdrawal Information not recorded | 8427 | 9112 | 8872 | 3689 | 1812 | 6249 | 3020

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10Pn3+1-6W-6M/043 Group | 10Pn2+1-6W-6M/043 Group | Ctrl-6W-6M/043 Group | 10Pn7-11M/043 Group | Ctrl7-11M/043 Group | 10Pn12-18M/043 Group | Ctrl12-18M/043 Group | Total
Number analyzed (Participants) | 8427 | 9112 | 8872 | 3689 | 1812 | 6249 | 3020 | 41181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8427 | 9112 | 8872 | 3689 | 1812 | 6249 | 3020 | 41181
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4239 | 4399 | 4351 | NA — Gender characteristics were not recorded for this group | NA — Gender characteristics were not recorded for this group | NA — Gender characteristics were not recorded for this group | NA — Gender characteristics were not recorded for this group | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 4188 | 4713 | 4521 | NA — Gender characteristics were not recorded for this group | NA — Gender characteristics were not recorded for this group | NA — Gender characteristics were not recorded for this group | NA — Gender characteristics were not recorded for this group | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Person Year Rate as Regards Subjects With Culture-confirmed IPD Due to Any of the 10 Pneumococcal Vaccine Serotypes. In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course
Description: The PYAR (Person-Year Rate) as regards subjects with culture-confirmed invasive pneumococcal disease (IPD) due to any of the pneumococcal vaccine serotypes was tabulated (vaccine pneumococcal serotypes = serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F). PYAR was calculated as follows n (= number of subjects reported with a culture confirmed IPD) divided by T (= sum of follow-up period expressed in years) (per 1000) as well as the corresponding 95% confidence interval (CI), calculated as a 2-sided profile log-likelihood ratio 95% CI using a classical log linear Poisson regression with strata.
Time Frame: Period of follow-up was any time after the administration of first vaccine dose till the end of the blinded invasive disease (ID) Follow-up period (The blinded ID Follow-up period lasted at least 30 months)
Population: The analysis was performed on the Infant Vaccinated cohort, which included all vaccinated,subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age and assigned to a 3-dose primary vaccination course.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Groups:
- 10Pn3+1-6W-6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) and 10PN-PDDIT-053 (NCT00839254 - EUDRACT 2008- 006551-51) (i.e. 1846 subjects) studies, pooled, and aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule). Refer to group description for 10Pn3+1-6W-6M/043 Group for vaccine specifics and administration route in this group.
- Ctrl-6W-6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) (i.e. 1329 subjects) studies, pooled, and aged 6 weeks to 6 months at enrolment. Subjects received the Engerix B vaccine (called also HBV vaccine) according to either a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule), or according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). Refer to group description for Ctrl6W-6M/043 Group for vaccine specifics and administration route in this group.
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10201
Participants per 1000 person-years | 0.000 [0.000 to 0.172] | 0.564 [0.291 to 0.984]
Statistical Analysis 1: Comparison: 10Pn3+1-6W-6M/043+053 Group vs Ctrl-6W-6M/043+053 Group; Analysis aimed at providing an estimate of vaccine effectiveness (VE) at preventing culture-confirmed IPD by comparing PYARs between groups taking into account the following parameters: T, n, n+ (number of clusters with at least one event culture-confirmed ID), and n/T. VE of the 10Pn vaccine in preventing culture-confirmed IPD due to the 10 vaccine serotypes was demonstrated if the 2-sided p-value calculated for the null hypothesis H0 =(vaccine-type [VT] IPD VE = 0%) was lower than (<) 5%; Test type: Superiority — VE (defined as 1 minus Relative Risk (RR)) was calculated by comparing numbers of culture-confirmed IPD. The number of subjects with IPD in each cluster was compared between groups (10PN3+1 vs Control). This comparison was done using a negative binomial log-linear model with correction for dispersion group- and cluster- related effect; p < 0.0001, Regression, Linear — P-value was calculated using a classical log linear Poisson regression with strata, without taking into account the multiplicity of the endpoints; VE (1-RR) = 100, 95% CI 2-sided [82.8 to 100]

2. Primary Outcome: Person Year Rate as Regards Subjects With Culture-confirmed IPD Due to Any of the 10 Pneumococcal Vaccine Serotypes. In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The analysis was performed on the Infant Vaccinated cohort, which included all vaccinated subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age and assigned to a 2-dose primary vaccination course.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Groups:
- 10Pn2+1-6W-6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) (i.e. 942 subjects) studies, pooled, and aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). Refer to group description for 10Pn2+1-6W-6M/043 Group for vaccine specifics and administration route in this group.
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10201
Participants per 1000 person-years | 0.048 [0.001 to 0.270] | 0.564 [0.291 to 0.984]
Statistical Analysis 1: Comparison: 10Pn2+1-6W-6M/043+053 Group vs Ctrl-6W-6M/043+053 Group; Analysis aimed at providing an estimate of vaccine effectiveness (VE) at preventing culture-confirmed IPD by comparing PYARs between groups taking into account the following parameters: T, n, n+ (number of clusters with at least one event culture-confirmed ID), and n/T. VE of the 10Pn vaccine in preventing culture-confirmed IPD due to the 10 vaccine serotypes was demonstrated if the 2-sided p-value calculated for the null hypothesis H0 = (vaccine-type [VT] IPD VE = 0%) was lower than (<) 5%; Test type: Superiority — VE (defined as 1 minus Relative Risk (RR)) was calculated by comparing numbers of culture-confirmed IPD. The number of subjects with IPD in each cluster was compared between groups (10PN2+1vsControl). This comparison was done using a negative binomial log-linear model with correction for dispersion group- and cluster- related effect; p = 0.0009, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; VE (1-RR) = 91.8, 95% CI 2-sided [58.3 to 99.6]

3. Secondary Outcome: Person Year Rate in the Prevention of Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course (Till End of Blinded ID FU Period)
Description: The PYAR (Person-Year Rate) was calculated as follows n (= number of subjects reported with a culture confirmed IPD) divided by T (= sum of follow-up period expressed in years) (per 1000) as well as the corresponding 95% confidence interval (CI), calculated as a 2-sided profile log- likelihood ratio 95% CI using a classical log linear Poisson regression with strata.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10201
Participants per 1000 person-years
  Culture confirmed ID | 0.093 [0.011 to 0.336] | 0.845 [0.501 to 1.336]
  Pneumococcal invasive disease (IPD) | 0.000 [0.000 to 0.172] | 0.657 [0.359 to 1.103]
  Serotype 4 | 0.000 [0.000 to 0.172] | 0.000 [0.000 to 0.173]
  Serotype 6B | 0.000 [0.000 to 0.172] | 0.235 [0.076 to 0.548]
  Serotype 7F | 0.000 [0.000 to 0.172] | 0.000 [0.000 to 0.173]
  Serotype 14 | 0.000 [0.000 to 0.172] | 0.188 [0.051 to 0.481]
  Serotype 18C | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Serotype 19F | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Serotype 23F | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Cross-reactive serotypes | 0.000 [0.000 to 0.172] | 0.094 [0.011 to 0.339]
  Serotype 6A | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Serotype 19A | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Other pneumococcal serotypes | 0.000 [0.000 to 0.172] | 0.000 [0.000 to 0.173]
  Serotype 3 | 0.000 [0.000 to 0.172] | 0.000 [0.000 to 0.173]
  Serotype 15C | 0.000 [0.000 to 0.172] | 0.000 [0.000 to 0.173]
  H. influenzae ID | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Non-typeable (NTHI) | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]
  Other bacteria | 0.093 [0.011 to 0.336] | 0.188 [0.051 to 0.481]
  Neisseria meningitidis | 0.093 [0.011 to 0.336] | 0.047 [0.001 to 0.262]
  Streptococcus pyogenes | 0.000 [0.000 to 0.172] | 0.094 [0.011 to 0.339]
  Moraxella catarrhalis | 0.000 [0.000 to 0.172] | 0.047 [0.001 to 0.262]

4. Secondary Outcome: Person Year Rate in the Prevention of Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course (Till End of Blinded ID FU Period)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10201
Participants per 1000 person-years
  Culture confirmed ID | 0.194 [0.053 to 0.496] | 0.845 [0.501 to 1.336]
  Pneumococcal invasive disease (IPD) | 0.097 [0.012 to 0.350] | 0.657 [0.359 to 1.103]
  Vaccine serotypes (vaccine type-IPD) | 0.048 [0.001 to 0.270] | 0.564 [0.291 to 0.984]
  Serotype 4 | 0.000 [0.000 to 0.179] | 0.000 [0.000 to 0.173]
  Serotype 6B | 0.000 [0.000 to 0.179] | 0.235 [0.076 to 0.548]
  Serotype 7F | 0.048 [0.001 to 0.270] | 0.000 [0.000 to 0.173]
  Serotype 14 | 0.000 [0.000 to 0.179] | 0.188 [0.051 to 0.481]
  Serotype 18C | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]
  Serotype 19F | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]
  Serotype 23F | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]
  Cross-reactive serotypes | 0.000 [0.000 to 0.179] | 0.094 [0.011 to 0.339]
  Serotype 6A | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]
  Serotype 19A | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]
  Other pneumococcal serotypes | 0.048 [0.001 to 0.270] | 0.000 [0.000 to 0.173]
  Serotype 3 | 0.048 [0.001 to 0.270] | 0.000 [0.000 to 0.173]
  Serotype 15C | 0.000 [0.000 to 0.179] | 0.000 [0.000 to 0.173]
  H. influenzae ID | 0.048 [0.001 to 0.270] | 0.047 [0.001 to 0.262]
  Non-typeable (NTHI) | 0.048 [0.001 to 0.270] | 0.047 [0.001 to 0.262]
  Other bacteria | 0.048 [0.001 to 0.270] | 0.188 [0.051 to 0.481]
  Neisseria meningitidis | 0.048 [0.001 to 0.270] | 0.047 [0.001 to 0.262]
  Streptococcus pyogenes | 0.000 [0.000 to 0.179] | 0.094 [0.001 to 0.339]
  Moraxella catarrhalis | 0.000 [0.000 to 0.179] | 0.047 [0.001 to 0.262]

5. Secondary Outcome: Person Year Rate in the Prevention of Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination in the 7-11 Months Schedule
Description: as for outcome 3
Time Frame: as for outcome 1
Population: The analysis was performed on the Catch-up Vaccinated cohort, which included all vaccinated subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with a 2-dose primary vaccination between 7 and 11 months of age.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Groups:
- 10Pn7-11M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) (i.e. 191 subjects) studies, pooled, and aged 7 to 11 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (11-17M Schedule). Refer to group description for 10Pn7-11M/043 Group for vaccine specifics and administration route in this group.
- Ctrl7-11M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) (i.e. 96 subjects) studies, pooled, and aged 7 to 11 months at enrolment. Subjects received the Engerix B (called also HBV) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (11-17M Schedule). Refer to group description for Ctrl7-11M/043 Group for vaccine specifics and administration route in this group.
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1908
Participants per 1000 person-years
  Culture confirmed ID | 0.000 [0.000 to 0.410] | 0.446 [0.054 to 1.612]
  Pneumococcal invasive disease (IPD) | 0.000 [0.000 to 0.410] | 0.446 [0.054 to 1.612]
  Vaccine serotypes (vaccine type-IPD) | 0.000 [0.000 to 0.410] | 0.446 [0.054 to 1.612]
  Serotype 4 | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 6B | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 7F | 0.000 [0.000 to 0.410] | 0.223 [0.006 to 1.243]
  Serotype 14 | 0.000 [0.000 to 0.410] | 0.223 [0.006 to 1.243]
  Serotype 18C | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 19F | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 23F | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Cross-reactive serotypes | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 6A | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 19A | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Other pneumococcal serotypes | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 3 | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Serotype 15C | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  H. influenzae ID | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Non-typeable (NTHI) | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Other bacteria | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]

6. Secondary Outcome: Person Year Rate in the Prevention of Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination in the 12-18 Months Schedule (+ Indirect Effects on the Unvaccinated Population)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: The analysis was performed on the Catch-up Vaccinated cohort, which included all vaccinated subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with a 2-dose primary vaccination between 12 and 18 months of age.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Groups:
- 10Pn12-18M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) (i.e. 286 subjects) studies, pooled, aged 12 to 18 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). Refer to group description for 10Pn12-18M/043 Group for vaccine specifics and administration route in this group.
- Ctrl12-18M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) and 10PN-PD-DIT-053 (NCT00839254 - EUDRACT 2008-006551-51) (i.e. 106 subjects) studies, pooled, and aged 12 to 18 months at enrolment. Subjects received the Havrix (called also HAV) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). Refer to group description for Ctrl12-18M/043 Group for vaccine specifics and administration route in this group.
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6535 | 3126
Participants per 1000 person-years
  Culture confirmed ID | 0.000 [0.000 to 0.240] | 0.674 [0.219 to 1.572]
  Pneumococcal invasive disease (IPD) | 0.000 [0.000 to 0.240] | 0.674 [0.219 to 1.572]
  Vaccine serotypes (vaccine type-IPD) | 0.000 [0.000 to 0.240] | 0.404 [0.083 to 1.181]
  Serotype 4 | 0.000 [0.000 to 0.240] | 0.135 [0.003 to 0.751]
  Serotype 6B | 0.000 [0.000 to 0.240] | 0.135 [0.003 to 0.751]
  Serotype 7F | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Serotype 14 | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Serotype 18C | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Serotype 19F | 0.000 [0.000 to 0.240] | 0.135 [0.0003 to 0.751]
  Serotype 23F | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Cross-reactive serotypes | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Serotype 6A | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Serotype 19A | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Other pneumococcal serotypes | 0.000 [0.000 to 0.240] | 0.269 [0.033 to 0.974]
  Serotype 3 | 0.000 [0.000 to 0.240] | 0.135 [0.003 to 0.751]
  Serotype 15C | 0.000 [0.000 to 0.240] | 0.135 [0.003 to 0.751]
  H. influenzae ID | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Non-typeable (NTHI) | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Other bacteria | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
Statistical Analysis 1: Comparison: 10Pn12-18M/043+053 Group; For indirect effectiveness analysis at preventing Culture-confirmed IPD (any serotype), number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any 10PN-PD-DIT vaccine - age stratum schedules); Test type: Other — In 5 to 99+ Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a classical log linear Poisson regression with strata). Total number of non-vaccinated persons = 2626735; Regression, Linear; Analysis performed on non-vaccinated persons, not enrolled in the study, but living in cluster areas in which study participants received vaccine; PYAR = 14.657, 95% CI 2-sided [13.229 to 16.197]
Statistical Analysis 2: Comparison: Ctrl12-18M/043+053 Group; For indirect effectiveness analysis at preventing Culture-confirmed IPD (any serotype), number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any control (HAV or HBV) vaccine - age stratum schedules); Test type: Other — In 5 to 99+ Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as the 95% CI (2-sided profile log-likelihood ratio 95% CI using a classical log linear Poisson regression with strata). Total number of non-vaccinated persons = 1354702; Regression, Linear; [statistical method as in outcome 6, analysis 1]; PYAR = 13.582, 95% CI 2-sided [11.691 to 15.693]
Statistical Analysis 3: Comparison: 10Pn12-18M/043+053 Group; For indirect effectiveness analysis at preventing Culture-confirmed IPD (vaccine serotype), number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any 10PN-PD-DIT vaccine - age stratum schedules); Test type: Other — [test comment as in outcome 6, analysis 1]; Regression, Linear; [statistical method as in outcome 6, analysis 1]; PYAR = 8.452, 95% CI 2-sided [7.376 to 9.639]
Statistical Analysis 4: Comparison: Ctrl12-18M/043+053 Group; For indirect effectiveness analysis at preventing Culture-confirmed IPD (vaccine serotype), number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any control (HAV or HBV) vaccine - age stratum schedules); Test type: Other — [test comment as in outcome 6, analysis 2]; Regression, Linear; [statistical method as in outcome 6, analysis 1]; PYAR = 7.603, 95% CI 2-sided [6.206 to 9.221]
Statistical Analysis 5: Comparison: 10Pn12-18M/043+053 Group; For indirect effectiveness analysis at preventing Culture-confirmed IPD (vaccine related), number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any 10PN-PD-DIT vaccine - age stratum schedules); Test type: Other — [test comment as in outcome 6, analysis 1]; Regression, Linear; [statistical method as in outcome 6, analysis 1]; PYAR = 1.637, 95% CI 2-sided [1.185 to 2.205]
Statistical Analysis 6: Comparison: Ctrl12-18M/043+053 Group; For indirect effectiveness analysis at preventing Culture-confirmed IPD (vaccine related), number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any control (HAV or HBV) vaccine - age stratum schedules); Test type: Other — [test comment as in outcome 6, analysis 2]; Regression, Linear; [statistical method as in outcome 6, analysis 1]; PYAR = 1.845, 95% CI 2-sided [1.194 to 2.724]
Statistical Analysis 7: Comparison: 10Pn12-18M/043+053 Group; For indirect effectiveness analysis at preventing Culture-confirmed IPD (non-vaccine & non-vaccine related), number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any 10PN-PD-DIT vaccine - age stratum schedules); Test type: Other — In 5 to 99+ Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as . 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons = 2626735; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 3.997, 95% CI 2-sided [3.269 to 4.839]
Statistical Analysis 8: Comparison: Ctrl12-18M/043+053 Group; For indirect effectiveness analysis at preventing Culture-confirmed IPD (non-vaccine & non-vaccine related), number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any control (HAV or HBV) vaccine - age stratum schedules); Test type: Other — In 5 to 99+ Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as the 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons = 1354702; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 3.322, 95% CI 2-sided [2.423 to 4.445]
Statistical Analysis 9: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 6, analysis 1]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =2636783; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 14.487, 95% CI 2-sided [13.071 to 16.015]
Statistical Analysis 10: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 6, analysis 2]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as the 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =1360966; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 13.740, 95% CI 2-sided [11.841 to 15.857]
Statistical Analysis 11: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 6, analysis 3]; Test type: Other — [test comment as in outcome 6, analysis 9]; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 7.813, 95% CI 2-sided [6.782 to 8.955]
Statistical Analysis 12: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 6, analysis 4]; Test type: Other — [test comment as in outcome 6, analysis 10]; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 7.789, 95% CI 2-sided [6.377 to 9.420]
Statistical Analysis 13: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 6, analysis 5]; Test type: Other — [test comment as in outcome 6, analysis 9]; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 2.313, 95% CI 2-sided [1.770 to 2.972]
Statistical Analysis 14: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 6, analysis 6]; Test type: Other — [test comment as in outcome 6, analysis 10]; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 1.984, 95% CI 2-sided [1.307 to 2.886]
Statistical Analysis 15: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 6, analysis 7]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model without strata). Total number of non-vaccinated persons =2636783; Negative Binomial model without strata; [statistical method as in outcome 6, analysis 1]; PYAR = 4.172, 95% CI 2-sided [3.429 to 5.028]
Statistical Analysis 16: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 6, analysis 8]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as the 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model without strata). Total number of non-vaccinated persons =1360966; Negative Binomial model without strata; [statistical method as in outcome 6, analysis 1]; PYAR = 3.968, 95% CI 2-sided [2.981 to 5.177]
Statistical Analysis 17: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 6, analysis 1]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =2654010; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 14.017, 95% CI 2-sided [12.628 to 15.516]
Statistical Analysis 18: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 6, analysis 2]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as the 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =1367343; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 15.066, 95% CI 2-sided [13.079 to 17.269]
Statistical Analysis 19: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 6, analysis 3]; Test type: Other — [test comment as in outcome 6, analysis 17]; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 5.916, 95% CI 2-sided [5.026 to 6.917]
Statistical Analysis 20: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 6, analysis 4]; Test type: Other — [test comment as in outcome 6, analysis 18]; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 8.557, 95% CI 2-sided [7.077 to 10.255]
Statistical Analysis 21: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 6, analysis 5]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a classical log linear Poisson regression with strata). Total number of non-vaccinated persons =2654010; Regression, Linear; [statistical method as in outcome 6, analysis 1]; PYAR = 2.977, 95% CI 2-sided [2.357 to 3.710]
Statistical Analysis 22: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 6, analysis 6]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with a culture confirmed IPD divided by sum of follow-up period expressed in years (per 100000), as well as the 95% CI (2-sided profile log-likelihood ratio 95% CI using a classical log linear Poisson regression with strata). Total number of non-vaccinated persons =1367343; Regression, Linear; [statistical method as in outcome 6, analysis 1]; PYAR = 2.048, 95% CI 2-sided [1.361 to 2.960]
Statistical Analysis 23: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 6, analysis 7]; Test type: Other — [test comment as in outcome 6, analysis 17]; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 5.011, 95% CI 2-sided [4.196 to 5.939]
Statistical Analysis 24: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 6, analysis 8]; Test type: Other — [test comment as in outcome 6, analysis 18]; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 4.315, 95% CI 2-sided [3.285 to 5.566]

7. Secondary Outcome: Person Year Rate in the Prevention of Probable Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course
Description: The PYAR (Person-Year Rate) was calculated as follows n (= number of subjects reported with a probable or culture confirmed ID) divided by T (= sum of follow-up period expressed in years) (per 1000) as well as the corresponding 95% confidence interval (CI), calculated as a 2-sided profile log-likelihood ratio 95% CI using a classical log linear Poisson regression with strata.
Time Frame: as for outcome 1
Population: The analysis was performed on the Infant Vaccinated cohort, which included all vaccinated subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age and assigned to a 3-dose primary vaccination course.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10201
Participants per 1000 person-years
  Probable cases of IPD | 0.000 [0.000 to 0.172] | 0.141 [0.029 to 0.412]
  Confirmed or probable cases of IPD | 0.000 [0.000 to 0.172] | 0.798 [0.465 to 1.278]

8. Secondary Outcome: Person Year Rate in the Prevention of Probable or Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course
Description: as for outcome 7
Time Frame: as for outcome 1
Population: The analysis was performed on the Infant Vaccinated cohort, all vaccinated subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age and assigned to a 2-dose primary vaccination course.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10201
Participants per 1000 person-years
  Probable cases of IPD | 0.000 [0.000 to 0.179] | 0.141 [0.029 to 0.412]
  Confirmed or probable cases of IPD | 0.097 [0.012 to 0.350] | 0.798 [0.465 to 1.278]

9. Secondary Outcome: Person Year Rate in the Prevention of Probable or Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination in the 7-11 Months Schedule
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1908
Participants per 1000 person-years
  Probable cases of IPD | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.823]
  Confirmed or probable cases of IPD | 0.000 [0.000 to 0.410] | 0.446 [0.054 to 1.612]

10. Secondary Outcome: Person Year Rate in the Prevention of Probable or Culture-confirmed Invasive Disease (ID)- In Children Starting Vaccination in the 12-18 Months Schedule (+ Indirect Effects on the Unvaccinated Population)
Description: The PYAR (Person-Year Rate) was calculated as follows n (= number of subjects reported with a probable or culture confirmed ID) divided by T (= sum of follow-up period expressed in years) (per 1000) as well as the corresponding 95% confidence interval (CI), calculated as a 2-sided profile log-likelihood ratio 95% CI using a classical log linear Poisson regression with strata. Data were not collected regarding indirect effects.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6535 | 3126
Participants per 1000 person-years
  Probable cases of IPD | 0.000 [0.000 to 0.240] | 0.000 [0.000 to 0.497]
  Confirmed or probable cases of IPD | 0.000 [0.000 to 0.240] | 0.674 [0.219 to 1.572]

11. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course
Description: PYAR was calculated: n (=number of subjects with hospital-diagnosed pneumonia) divided by T (=sum of follow-up (FU) period expressed in years) (per 1000) with 95% CI (2-sided profile log-likelihood ratio 95% CI-classical log linear Poisson regression with strata). FU period considered as period between Dose 1 administration and cut-off date of 31 December 2011. Hospital-diagnosed pneumonia (HDP) cases identified based on hospital discharge diagnosis using international Classification of Disease (ICD)-10 diagnosis codes: J10.0 (Influenza with HDP, other influenza virus identified), J11.0 (Influenza with HDP, virus not identified), J12 (Viral HDP, not elsewhere classified), J13 (HDP due to Sp.), J14 (for HDP due to Hi.), J15 (all HDP, not elsewhere classified), J16 (HDP due to other infectious organisms, not elsewhere classified), J17 (HDP in diseases classified elsewhere), J18 (HDP organism unspecified), J85.1 (Abscess of lung with HDP), and J86 (Pyothorax including empyema).
Time Frame: Period of follow-up was any time after the administration of first vaccine dose till the end date of the follow-up (31 December 2011) - FU mean time=24 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10200
Participants per 1000 person-years | 10.131 [8.804 to 11.601] | 13.854 [12.287 to 15.566]

12. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course
Description: PYAR was calculated: n (= number of subjects with hospital-diagnosed pneumonia) divided by T (= sum of follow-up (FU) period expressed in years) (per 1000) with 95% CI (2-sided profile log-likelihood ratio 95% CI-classical log linear Poisson regression with strata). FU period considered as period between Dose 1 administration and cut-off date of 31 December 2011. Hospital-diagnosed pneumonia (HDP) cases identified based on hospital discharge diagnosis using international Classification of Disease (ICD)-10 diagnosis codes: J10.0 (Influenza with HDP, other influenza virus identified), J11.0 (Influenza with HDP, virus not identified), J12 (Viral HDP, not elsewhere classified), J13 (HDP due to Sp.), J14 (for HDP due to Hi.), J15 (all HDP, not elsewhere classified), J16 (HDP due to other infectious organisms, not elsewhere classified), J17 (HDP in diseases classified elsewhere), J18 (HDP organism unspecified), J85.1 (Abscess of lung with HDP), and J86 (Pyothorax including empyema).
Time Frame: as for outcome 11
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10200
Participants per 1000 person-years | 10.155 [8.800 to 11.660] | 13.854 [12.287 to 15.566]

13. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia- In Children Starting Vaccination in the 7-11 Months Schedule
Description: as for outcome 12
Time Frame: Period of follow-up was any time after the administration of first vaccine dose till the end date of the follow-up (31 December 2011) - FU mean time=27 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1907
Participants per 1000 person-years | 10.263 [8.242 to 12.630] | 15.752 [12.232 to 19.970]

14. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia - In Children Starting Vaccination in the 12-18 Months Schedule (+ Indirect Effects on the Unvaccinated Population)
Description: as for outcome 12
Time Frame: as for outcome 13
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6534 | 3126
Participants per 1000 person-years | 9.322 [7.832 to 11.013] | 11.739 [9.363 to 14.533]
Statistical Analysis 1: Comparison: 10Pn12-18M/043+053 Group; For indirect effectiveness analysis at preventing Hospital-diagnosed Pneumonia, number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any 10PN-PD-DIT vaccine - age stratum schedules); Test type: Other — In 5 to 99+ Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with a Hospital-diagnosed Pneumonia divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =2626735; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 9.218, 95% CI 2-sided [9.103 to 9.335]
Statistical Analysis 2: Comparison: Ctrl12-18M/043+053 Group; For indirect effectiveness analysis at preventing Hospital-diagnosed Pneumonia, number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any control (HAV or HBV) vaccine - age stratum schedules); Test type: Other — In 5 to 99+ Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with a Hospital-diagnosed Pneumonia divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =1354702; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 9.212, 95% CI 2-sided [9.052 to 9.375]
Statistical Analysis 3: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 14, analysis 1]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with a Hospital-diagnosed Pneumonia divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =2636783; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 10.500, 95% CI 2-sided [10.378 to 10.624]
Statistical Analysis 4: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 14, analysis 2]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with a Hospital-diagnosed Pneumonia divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =1360966; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 10.429, 95% CI 2-sided [10.259 to 10.601]
Statistical Analysis 5: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 14, analysis 1]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with a Hospital-diagnosed Pneumonia divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =2654010; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 10.118, 95% CI 2-sided [9.997 to 10.239]
Statistical Analysis 6: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 14, analysis 2]; Test type: Other — In 5 to 99+ Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with a Hospital-diagnosed Pneumonia divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =1367343; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 9.921, 95% CI 2-sided [9.755 to 10.088]

15. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia With Chest X-ray (CXR) Reading According to WHO Criteria- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course
Description: PYAR was calculated: n (= number of subjects with hospital-diagnosed pneumonia [HDP]) divided by T (= sum of follow-up (FU) period expressed in years) (per 1000) with 95% CI (2-sided profile log-likelihood ratio 95% CI-classical log linear Poisson regression with strata for non-consolidated HDP and without strata for consolidated HDP). FU period considered as period between Dose 1 administration and cut-off date of 31 December 2011. CXR HDP was defined as a HDP case with the presence of abnormal pulmonary infiltrates on the CXR as per independent review panel judgement using WHO methodology. Abnormal pulmonary infiltrates could be either with (Consolidated HDP) or without (Non-consolidated HDP) alveolar consolidation/pleural effusion. New cases of HDP and CXR HDP were based on a 30-day rule, i.e. a new episode was considered if at least a 30-day interval elapsed from the onset of the previous episode.
Time Frame: as for outcome 11
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10200
Participants per 1000 person-years
  Consolidated pneumonia | 2.181 [1.591 to 2.919] | 3.965 [3.149 to 4.929]
  Non-consolidated pneumonia | 2.908 [2.219 to 3.744] | 2.937 [2.241 to 3.781]
  Consolidated or non- consolidated pneumonia | 5.090 [4.163 to 6.161] | 6.903 [5.810 to 8.141]

16. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia With CXR Reading According to WHO Criteria - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course
Description: as for outcome 15
Time Frame: as for outcome 11
Population: The analysis was performed on the Infant Vaccinated cohort, which included all vaccinated,subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age and assigned to a 2-dose primary vaccination course.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10200
Participants per 1000 person-years
  Consolidated pneumonia | 2.273 [1.658 to 3.042] | 3.965 [3.149 to 4.929]
  Non-consolidated pneumonia | 2.627 [1.962 to 3.445] | 2.937 [2.241 to 3.781]
  Consolidated or non- consolidated pneumonia | 4.901 [3.974 to 5.978] | 6.903 [5.810 to 8.141]

17. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia With CXR Reading According to WHO Criteria - In Children Starting Vaccination in the 7-11 Months Schedule
Description: as for outcome 15
Time Frame: as for outcome 13
Population: The analysis was performed on the Catch-up Vaccinated cohort, which included all vaccinated,subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with a 2-dose primary vaccination between 7 and 11 months of age.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1907
Participants per 1000 person-years
  Consolidated pneumonia | 1.960 [1.142 to 3.139] | 4.401 [2.650 to 6.873]
  Non-consolidated pneumonia | 3.344 [2.240 to 4.803] | 4.865 [3.011 to 7.436]
  Consolidated or non- consolidated pneumonia | 5.305 [3.884 to 7.076] | 9.266 [6.620 to 12.618]

18. Secondary Outcome: Person Year Rate in Reducing Hospital-diagnosed Pneumonia With CXR Reading According to WHO Criteria - In Children Starting Vaccination in the 12-18 Months Schedule
Description: as for outcome 15
Time Frame: as for outcome 13
Population: The analysis was performed on the Catch-up Vaccinated cohort, which included all vaccinated,subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with a 2-dose primary vaccination between 12 and 18 months of age.
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6534 | 3126
Participants per 1000 person-years
  Consolidated pneumonia | 1.824 [1.202 to 2.654] | 3.494 [2.261 to 5.157]
  Non-consolidated pneumonia | 2.837 [2.045 to 3.835] | 2.935 [1.817 to 4.486]
  Consolidated or non- consolidated pneumonia | 4.661 [3.626 to 5.899] | 6.428 [4.706 to 8.574]

19. Secondary Outcome: Person Year Rate in Prevention of All Tympanostomy Tube Placements- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course
Description: PYAR was calculated: n (= number of subjects with tympanostomy tube placement[TTP]) divided by T (= sum of follow-up (FU) period expressed in years) (per 1000) with 95% CI (2-sided profile log-likelihood ratio 95% CI-classical log linear Poisson regression with strata). FU period considered as period between Dose 1 administration and cut-off date of 31 December 2011. A TTP episode was defined as a TTP episode classified under the DCA 20 code in the Finnish National Institute of Health and Welfare (THL) and Social Insurance Institution of Finland (KELA) registers, using the Nordic Centre for Classifications in Health Care (NOMESCO) Classification of Surgical Procedures (NCSP), version 1.12 from January 2008, and could refer to either an unilateral or a bilateral TTP procedure. New episodes of TTP defined according to a 30-day rule meaning that a new episode was considered if at least 30-day interval elapsed from the onset of the previous episode.
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10200
Participants per 1000 person-years | 68.735 [65.203 to 72.408] | 79.504 [75.683 to 83.467]

20. Secondary Outcome: Person Year Rate in Prevention of All Tympanostomy Tube Placements - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course
Description: as for outcome 19
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10200
Participants per 1000 person-years | 66.083 [62.550 to 69.764] | 79.504 [75.683 to 83.467]

21. Secondary Outcome: Person Year Rate in Prevention of All Tympanostomy Tube Placements - In Children Starting Vaccination in the 7-11 Months Schedule
Description: as for outcome 19
Time Frame: as for outcome 13
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1907
Participants per 1000 person-years | 68.153 [62.769 to 73.876] | 79.920 [71.708 to 88.814]

22. Secondary Outcome: Person Year Rate in Prevention of All Tympanostomy Tube Placements - In Children Starting Vaccination in the 12-18 Months Schedule (+ Indirect Effects on the Unvaccinated Population)
Description: as for outcome 19
Time Frame: as for outcome 13
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6534 | 3126
Participants per 1000 person-years | 56.809 [53.034 to 60.782] | 58.973 [53.480 to 64.877]
Statistical Analysis 1: Comparison: 10Pn12-18M/043+053 Group; For indirect effectiveness analysis at preventing Tympanostomy Tube Placements, number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any 10PN-PD-DIT vaccine - age stratum schedules); Test type: Other — In 0 to 7 Years Old Population, in Year 2009, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with Tympanostomy Tube Placement divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =229978; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 22.624, 95% CI 2-sided [22.020 to 23.240]
Statistical Analysis 2: Comparison: Ctrl12-18M/043+053 Group; For indirect effectiveness analysis at preventing Tympanostomy Tube Placements, number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any control (HAV or HBV) vaccine - age stratum schedules); Test type: Other — In 0 to 7 Years Old Population, in Year 2009, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with Tympanostomy Tube Placement divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =120190; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 22.747, 95% CI 2-sided [21.912 to 23.606]
Statistical Analysis 3: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 22, analysis 1]; Test type: Other — In 0 to 7 Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with Tympanostomy Tube Placement divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =214181; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 24.503, 95% CI 2-sided [23.852 to 25.166]
Statistical Analysis 4: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 22, analysis 2]; Test type: Other — In 0 to 7 Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with Tympanostomy Tube Placement divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =112060; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 26.236, 95% CI 2-sided [25.308 to 27.189]
Statistical Analysis 5: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 22, analysis 1]; Test type: Other — In 0 to 7 Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with Tympanostomy Tube Placement divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =211914; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 27.502, 95% CI 2-sided [26.810 to 28.207]
Statistical Analysis 6: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 22, analysis 2]; Test type: Other — In 0 to 7 Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with Tympanostomy Tube Placement divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =111071; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 26.100, 95% CI [25.171 to 27.055]
Statistical Analysis 7: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 22, analysis 1]; Test type: Other — In 0 to 7 Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with Tympanostomy Tube Placement divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =213913; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 28.661, 95% CI 2-sided [27.958 to 29.377]
Statistical Analysis 8: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 22, analysis 2]; Test type: Other — In 0 to 7 Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with Tympanostomy Tube Placement divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =111414; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 29.835, 95% CI 2-sided [28.843 to 30.850]

23. Secondary Outcome: Person Year Rate in Prevention of All Antimicrobial Prescriptions- In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course
Description: PYAR was calculated: n (= number of subjects with antimicrobial prescriptions (APs)) divided by T (= sum of follow-up (FU) period expressed in years) (per 1000) with 95% CI (2-sided profile log-likelihood ratio 95% CI-classical log linear Poisson regression with strata). FU period considered as period between Dose 1 administration and cut-off date of 31 December 2011. An APs episode was an episode of APs to an infant/child falling under following Anatomic Therapeutic Chemical [ATC] codes: J01 (APs) and following codes for AP usually recommended for otitis media (OM) and respiratory tract infections (RTI). "For OM and RTI" category corresponds to following definition: APs for antibacterial usually recommended for OM and RTI (ATC codes: J01CA04, J01CR02, J01CE02, J01DC02, J01DC04, J01EE02, J01FA09 and J01FA10). New episodes of APs were analyzed according to a 2-day rule meaning new episode considered if at least 2 day interval elapsed from the onset of the previous episode.
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10273 | 10200
Participants per 1000 person-years
  Antimicrobial prescriptions (ATC code J01) | 1592.585 [1575.411 to 1609.901] | 1706.194 [1688.328 to 1724.202]
  For otitis media and respiratory infections | 1451.141 [1434.749 to 1467.674] | 1565.692 [1548.579 to 1582.947]

24. Secondary Outcome: Person Year Rate in Prevention of All Antimicrobial Prescriptions - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course
Description: as for outcome 23
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10054 | 10200
Participants per 1000 person-years
  Antimicrobial prescriptions (ATC code J01) | 1552.493 [1535.183 to 1569.950] | 1706.194 [1688.328 to 1724.202]
  For otitis media and respiratory infections | 1415.983 [1399.453 to 1432.659] | 1565.692 [1548.579 to 1582.947]

25. Secondary Outcome: Person Year Rate in Prevention of All Antimicrobial Prescriptions - In Children Starting Vaccination in the 7-11 Months Schedule
Description: as for outcome 23
Time Frame: as for outcome 13
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group
Number analyzed (Participants) | 3880 | 1907
Participants per 1000 person-years
  Antimicrobial prescriptions (ATC code J01) | 1536.618 [1510.637 to 1562.934] | 1649.360 [1611.269 to 1688.124]
  For otitis media and respiratory infections | 1390.856 [1366.143 to 1415.903] | 1499.713 [1463.401 to 1536.698]

26. Secondary Outcome: Person Year Rate in Prevention of All Antimicrobial Prescriptions - In Children Starting Vaccination in the 12-18 Months Schedule (+ Indirect Effects on the Unvaccinated Population)
Description: as for outcome 23
Time Frame: as for outcome 13
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 6534 | 3126
Participants per 1000 person-years
  Antimicrobial prescriptions (ATC code J01) | 1315.936 [1297.521 to 1334.547] | 1421.774 [1394.280 to 1449.675]
  For otitis media and respiratory infections | 1177.729 [1160.312 to 1195.343] | 1271.268 [1245.277 to 1297.665]
Statistical Analysis 1: Comparison: 10Pn12-18M/043+053 Group; For indirect effectiveness analysis at preventing Antimicrobial Prescriptions, number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any 10PN-PD-DIT vaccine - age stratum schedules); Test type: Other — In 0 to 7 Years Old Population, in Year 2009, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =229978; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 816.813, 95% CI 2-sided [815.226 to 818.392]
Statistical Analysis 2: Comparison: Ctrl12-18M/043+053 Group; For indirect effectiveness analysis at preventing Antimicrobial Prescriptions, number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any control (HAV or HBV) vaccine - age stratum schedules); Test type: Other — In 0 to 7 Years Old Population, in Year 2009, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =120190; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 841.176, 95% CI 2-sided [839.098 to 843.239]
Statistical Analysis 3: Comparison: 10Pn12-18M/043+053 Group; For indirect effectiveness analysis at preventing Antimicrobial Prescriptions recommended for Acute Otitis Media (AOM)/Respiratory Tract Infections (RTI), number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any 10PN-PD-DIT vaccine - age stratum schedules); Test type: Other — In 0 to 7 Years Old Population, in Year 2009, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with recommended Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =229978; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 702.245, 95% CI 2-sided [700.372 to 704.114]
Statistical Analysis 4: Comparison: Ctrl12-18M/043+053 Group; For indirect effectiveness analysis at preventing Antimicrobial Prescriptions recommended for AOM/RTI, number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any control (HAV or HBV) vaccine - age stratum schedules); Test type: Other — In 0 to 7 Years Old Population, in Year 2009, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with recommended Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =120190; negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 720.900, 95% CI 2-sided [718.355 to 723.435]
Statistical Analysis 5: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 26, analysis 1]; Test type: Other — In 0 to 7 Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =214181; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 929.844, 95% CI 2-sided [928.755 to 930.923]
Statistical Analysis 6: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 26, analysis 2]; Test type: Other — In 0 to 7 Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =112060; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 953.025, 95% CI 2-sided [951.770 to 954.257]
Statistical Analysis 7: Comparison: 10Pn12-18M/043+053 Group; For indirect effectiveness analysis at preventing Antimicrobial Prescriptions recommended for AOM/RTI, number of events in the unvaccinated cohort, which occurred around 6 months or more after study start was compared with treated group numbers (applicable to any 10PN-PD-DIT vaccine - age stratum schedules); Test type: Other — In 0 to 7 Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with recommended Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =214181; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 804.703, 95% CI 2-sided [803.017 to 806.380]
Statistical Analysis 8: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 26, analysis 4]; Test type: Other — In 0 to 7 Years Old Population, in Year 2010, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with recommended Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =112060; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 818.660, 95% CI 2-sided [816.391 to 820.912]
Statistical Analysis 9: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 26, analysis 1]; Test type: Other — In 0 to 7 Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =211914; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 916.079, 95% CI 2-sided [914.891 to 917.256]
Statistical Analysis 10: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 26, analysis 2]; Test type: Other — In 0 to 7 Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =111071; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 928.568, 95% CI 2-sided [927.038 to 930.076]
Statistical Analysis 11: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 26, analysis 7]; Test type: Other — In 0 to 7 Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with recommended Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =211914; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 796.894, 95% CI [795.175 to 798.605]
Statistical Analysis 12: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 26, analysis 4]; Test type: Other — In 0 to 7 Years Old Population, in Year 2011, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with recommended Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =111071; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 803.918, 95% CI 2-sided [801.571 to 806.250]
Statistical Analysis 13: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 26, analysis 1]; Test type: Other — In 0 to 7 Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =213913; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 865.679, 95% CI 2-sided [864.227 to 867.121]
Statistical Analysis 14: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 26, analysis 2]; Test type: Other — In 0 to 7 Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =111414; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 871.749, 95% CI 2-sided [869.771 to 873.707]
Statistical Analysis 15: Comparison: 10Pn12-18M/043+053 Group; [analysis description as in outcome 26, analysis 7]; Test type: Other — In 0 to 7 Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received 10Pn-PD-DiT vaccine, PYAR was calculated (= number of subjects reported with recommended Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =213913; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 753.423, 95% CI 2-sided [751.591 to 755.249]
Statistical Analysis 16: Comparison: Ctrl12-18M/043+053 Group; [analysis description as in outcome 26, analysis 4]; Test type: Other — In 0 to 7 Years Old Population, in Year 2012, for Non-vaccinated persons living in study cluster areas, in which study participants received control vaccine, PYAR was calculated (= number of subjects reported with recommended Antimicrobial Prescriptions divided by sum of follow-up period expressed in years (per 1000), as well as 95% CI (2-sided profile log-likelihood ratio 95% CI using a Negative Binomial regression model with strata). Total number of non-vaccinated persons =111414; Negative Binomial model with strata; [statistical method as in outcome 6, analysis 1]; PYAR = 755.542, 95% CI 2-sided [753.008 to 758.064]

27. Secondary Outcome: Number of Subjects Classified by Antimicrobial Susceptiblity of IPD Isolates in Children Starting Vaccination Within 7 Months of Life and Assigned to a 2 or 3-dose Primary Vaccination Course
Description: Antimicrobial susceptibility classification of IPD isolates reported during IPD follow-up with percentages for each serotype for the following categories: S= susceptible; I = intermediate ; R = resistant; N = not available.
Time Frame: Period of follow-up was any time after the administration of first vaccine dose till the end date of the follow-up (31 December 2011) - mean FU time=24 months
Population: The analysis was performed on the Infant Vaccinated cohort, which included all vaccinated,subjects in the 10PN-PD-DIT-043 study and vaccinated subjects of 10PN-PD-DIT-053 study who contributed to the effectiveness analysis, with first dose of study vaccine below 7 months of age.
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 0 | 2 | 24
Participants
  Serotype-4 -Pencillin-S |  | 0 | 1
  Serotype-6A -Pencillin-S |  | 0 | 1
  Serotype-6B -Pencillin-I |  | 0 | 3
  Serotype-6B -Pencillin-R |  | 0 | 1
  Serotype-6B -Pencillin-S |  | 0 | 2
  Serotype-7F -Pencillin-S |  | 1 | 1
  Serotype-14 -Pencillin-I |  | 0 | 2
  Serotype-14 -Pencillin-R |  | 0 | 1
  Serotype-14 -Pencillin-S |  | 0 | 2
  Serotype-15C -Pencillin-S |  | 0 | 1
  Serotype-18C -Pencillin-S |  | 0 | 1
  Serotype-19A -Pencillin-I |  | 0 | 1
  Serotype-19F -Pencillin-I |  | 0 | 1
  Serotype-19F -Pencillin-S |  | 0 | 1
  Serotype-23F -Pencillin-S |  | 0 | 1
  Serotype-N -Pencillin-N |  | 1 | 4
  Serotype-4 -Erythromycin-S |  | 0 | 1
  Serotype-6A -Erythromycin-S |  | 0 | 1
  Serotype-6B -Erythromycin-R |  | 0 | 5
  Serotype-6B -Erythromycin-S |  | 0 | 1
  Serotype-7F -Erythromycin-S |  | 1 | 1
  Serotype-14 -Erythromycin-R |  | 0 | 4
  Serotype-14 -Erythromycin-S |  | 0 | 1
  Serotype-15C -Erythromycin-S |  | 0 | 1
  Serotype-18C -Erythromycin-S |  | 0 | 1
  Serotype-19A -Erythromycin-S |  | 0 | 1
  Serotype-19F -Erythromycin-R |  | 0 | 1
  Serotype-19F -Erythromycin-S |  | 0 | 1
  Serotype-23F -Erythromycin-S |  | 0 | 1
  Serotype-N -Erythromycin-N |  | 1 | 4
  Serotype-4 -Tetracyclin-S |  | 0 | 1
  Serotype-6A -Tetracyclin-S |  | 0 | 1
  Serotype-6B -Tetracyclin-R |  | 0 | 4
  Serotype-6B -Tetracyclin-S |  | 0 | 2
  Serotype-7F -Tetracyclin-S |  | 1 | 1
  Serotype-14 -Tetracyclin-S |  | 0 | 5
  Serotype-15C -Tetracyclin-S |  | 0 | 1
  Serotype-18C -Tetracyclin-S |  | 0 | 1
  Serotype-19A -Tetracyclin-S |  | 0 | 1
  Serotype-19F -Tetracyclin-R |  | 0 | 1
  Serotype-19F -Tetracyclin-S |  | 0 | 1
  Serotype-23F -Tetracyclin-S |  | 0 | 1
  Serotype-N -Tetracyclin-N |  | 1 | 4
  Serotype-4 -Levoffloxacin-S |  | 0 | 1
  Serotype-6A -Levoffloxacin-S |  | 0 | 1
  Serotype-6B -Levoffloxacin-S |  | 0 | 6
  Serotype-7F -Levoffloxacin-S |  | 1 | 1
  Serotype-14 -Levoffloxacin-S |  | 0 | 5
  Serotype-15C -Levoffloxacin-S |  | 0 | 1
  Serotype-18C -Levoffloxacin-S |  | 0 | 1
  Serotype-19A -Levoffloxacin-S |  | 0 | 1
  Serotype-19F -Levoffloxacin-S |  | 0 | 2
  Serotype-23F -Levoffloxacin-S |  | 0 | 1
  Serotype-N -Levoffloxacin-N |  | 1 | 4
  Serotype-4 -Ceftriaxone-S |  | 0 | 1
  Serotype-6A -Ceftriaxone-S |  | 0 | 1
  Serotype-6B -Ceftriaxone-S |  | 0 | 6
  Serotype-7F -Ceftriaxone-S |  | 1 | 1
  Serotype-14 -Ceftriaxone-I |  | 0 | 1
  Serotype-14 -Ceftriaxone-S |  | 0 | 4
  Serotype-15C -Ceftriaxone-S |  | 0 | 1
  Serotype-18C -Ceftriaxone-S |  | 0 | 1
  Serotype-19A -Ceftriaxone-S |  | 0 | 1
  Serotype-19F -Ceftriaxone-S |  | 0 | 2
  Serotype-23F -Ceftriaxone-S |  | 0 | 1
  Serotype-N -Ceftriaxone-N |  | 1 | 4
  Serotype-4 -Clindamycin-S |  | 0 | 1
  Serotype-6A -Clindamycin-S |  | 0 | 1
  Serotype-6B -Clindamycin-R |  | 0 | 4
  Serotype-6B -Clindamycin-S |  | 0 | 2
  Serotype-7F -Clindamycin-S |  | 1 | 1
  Serotype-14 -Clindamycin-N |  | 0 | 1
  Serotype-14 -Clindamycin-S |  | 0 | 4
  Serotype-15C -Clindamycin-S |  | 0 | 1
  Serotype-18C -Clindamycin-S |  | 0 | 1
  Serotype-19A -Clindamycin-S |  | 0 | 1
  Serotype-19F -Clindamycin-R |  | 0 | 1
  Serotype-19F -Clindamycin-S |  | 0 | 1
  Serotype-23F -Clindamycin-S |  | 0 | 1
  Serotype-N -Clindamycin-N |  | 1 | 4

28. Secondary Outcome: Number of Subjects With Lower Respiratory Tract Infections (LRTIs) (in a Subset of Subjects in Turku Area)
Description: Analysis of this outcome was performed in the Turku area. The number of subjects reporting at least one LRTI any time after the administration of the first vaccine dose was tabulated.
Time Frame: From the administration of the first vaccine dose till the end of the blinded invasive disease (ID) Follow-up period (at least 30 months)
Population: The analysis was performed in a subset of vaccinated subjects including all vaccinated subjects enrolled in the 10PN-PD-DIT-053 study in the Turku area and those vaccinated subjects enrolled in the 10PN-PD-DIT-043 study in the Turku area who agreed to take part in this assessment.
Measure: Count of Participants; unit: Participants
Groups:
- 10Pn2+1-6W-6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) and 10PN-PDDIT-053 (NCT00839254 - EUDRACT 2008- 006551-51) (i.e. 942 subjects) studies, pooled, and aged 6 weeks to 6 months at enrolment. Subjects received the Synflorix (called also 10Pn-PD-DiT, 10Pn or GSK1024850A) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks, followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). Refer to group description for 10Pn2+1-6W-6M/043 Group for vaccine specifics and administration route in this group.
- Ctrl-6W-6M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) and 10PN-PDDIT-053 (NCT00839254 - EUDRACT 2008- 006551-51) (i.e. 1329 subjects) studies, pooled, and aged 6 weeks to 6 months at enrolment. Subjects received the Engerix B vaccine (called also HBV vaccine) according to either a 3-dose primary vaccination schedule with an interval of at least 4 weeks between doses followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (3+1 Infant Schedule), or according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (2+1 Infant Schedule). Refer to group description for Ctrl6W-6M/043 Group for vaccine specifics and administration route in this group.
- Ctrl7-11M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) and 10PN-PDDIT-053 (NCT00839254 - EUDRACT 2008-006551-51) (i.e. 96 subjects) studies, pooled, and aged 7 to 11 months at enrolment. Subjects received the Engerix B (called also HBV) vaccine according to a 2-dose primary vaccination with an interval of at least 8 weeks followed by a booster dose of the same vaccine with an interval of preferably 6 months since the previous vaccine dose (minimum 4 months) (11-17M Schedule). Refer to group description for Ctrl7-11M/043 Group for vaccine specifics and administration route in this group.
- 10Pn12-18M/043+053 Group: Subjects in this group were subjects enrolled in the 10PN-PD-DIT-043 (NCT00861380 - EUDRACT 2008-005149-48) and 10PN-PDDIT-053 (NCT00839254 - EUDRACT 2008-006551-51) (i.e. 286 subjects) studies, pooled, aged 12 to 18 months at enrolment. Subjects received the Synflorix (called also 10Pn-PDDiT, 10Pn or GSK1024850A) vaccine according to a 2-dose vaccination with an interval of at least and preferably 6 months between doses (12-18M Schedule). Refer to group description for 10Pn12-18M/043 Group for vaccine specifics and administration route in this group.
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 243 | 190 | 171 | 31 | 22 | 62 | 48
Participants | 19 | 19 | 19 | 3 | 1 | 5 | 2

29. Secondary Outcome: Number of Subjects With Upper Respiratory Tract Infections (URTIs) (in a Subset of Subjects in Turku Area)
Description: Analysis of this outcome was performed in the Turku area. The number of subjects reporting at least one URTI any time after the administration of the first vaccine dose was tabulated.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 243 | 190 | 171 | 31 | 22 | 62 | 48
Participants | 158 | 124 | 94 | 14 | 15 | 27 | 19

30. Secondary Outcome: Number of Subjects With SAEs Reported During the Blinded Invasive Disease Phase, of the Study
Description: An event is defined as 'serious' when it meets one of the pre-defined outcomes described below: results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation; results in disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a study subject.
  Medical or scientific judgement should be exercised in deciding whether reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalisation but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These should also be considered serious.
Time Frame: For Month 0 till the end of the blinded ID Follow-Up, (at least 30 months from study start)
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/043 Group | 10Pn2+1-6W-6M/043 Group | Ctrl-6W-6M/043 Group | 10Pn7-11M/043 Group | Ctrl7-11M/043 Group | 10Pn12-18M/043 Group | Ctrl12-18M/043 Group
Number analyzed (Participants) | 8427 | 9112 | 8872 | 3689 | 1812 | 6249 | 3020
Participants | 6 | 7 | 8 | 3 | 2 | 2 | 2

31. Secondary Outcome: Number of Subjects Enrolled and Vaccinated in the 10PN-PD-DIT-043 and 10PN-PD-DIT-053 Study With Post-study SAEs Reported Via Passive Surveillance- Subjects Enrolled Aged 6 Weeks to 6 Months and 7 to 18 Months
Description: as for outcome 30
Time Frame: From the end of the blinded ID Follow-Up period(at least 30 months from study start) up to the end of 18-month period after study unblinding
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group | 10Pn7-11M/043+053 Group | Ctrl7-11M/043+053 Group | 10Pn12-18M/043+053 Group | Ctrl12-18M/043+053 Group
Number analyzed (Participants) | 10273 | 10054 | 10201 | 3880 | 1908 | 6535 | 3126
Participants | 1 | 2 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Culture-confirmed Invasive Disease (ID) Person Year Rate - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 3-dose Primary Vaccination Course Till End of LT FU Period
Description: The PYAR (Person-Year Rate) was calculated as follows n (= number of subjects reported with a culture confirmed IPD) divided by T (= sum of follow-up period expressed in years) (per 1000) as well as the corresponding 95% confidence interval (CI), calculated as a 2-sided profile log-likelihood ratio 95% CI using a classical log linear Poisson regression with strata.
Time Frame: Period of follow-up was any time after the administration of first vaccine dose till the end of the long-term Follow-up period (The Follow-up period lasted at least 77 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn3+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10272 | 10201
Participants per 1000 person-years
  Culture confirmed ID | 0.046 [0.013 to 0.118] | 0.268 [0.170 to 0.402]
  Pneumococcal invasive disease (IPD) | 0.023 [0.003 to 0.084] | 0.210 [0.124 to 0.331]
  Vaccine serotypes (vaccine type-IPD) | 0.0 [0.0 to 0.043] | 0.140 [0.072 to 0.244]
  Serotype 4 | 0.0 [0.0 to 0.043] | 0.0 [0.0 to 0.043]
  Serotype 6B | 0.0 [0.0 to 0.043] | 0.058 [0.019 to 0.136]
  Serotype 7F | 0.0 [0.0 to 0.043] | 0.0 [0.0 to 0.043]
  Serotype 14 | 0.0 [0.0 to 0.043] | 0.047 [0.013 to 0.119]
  Serotype 18C | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Serotype 19F | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Serotype 23F | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Cross-reactive serotypes | 0.012 [0.0 to 0.064] | 0.047 [0.013 to 0.119]
  Serotype 6A | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Serotype 19A | 0.012 [0.0 to 0.064] | 0.035 [0.007 to 0.102]
  Other pneumococcal serotypes | 0.012 [0.0 to 0.064] | 0.023 [0.003 to 0.084]
  Serotype 3 | 0.012 [0.0 to 0.064] | 0.012 [0.0 to 0.065]
  Serotype 12F | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Serotype 15C | 0.0 [0.0 to 0.043] | 0.0 [0.0 to 0.043]
  H. influenzae ID | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Non-typeable (NTHI) | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]
  Other bacteria | 0.023 [0.003 to 0.084] | 0.058 [0.019 to 0.136]
  Neisseria meningitidis | 0.023 [0.003 to 0.084] | 0.023 [0.003 to 0.084]
  Streptococcus pyogenes | 0.0 [0.0 to 0.043] | 0.023 [0.003 to 0.084]
  Moraxella catarrhalis | 0.0 [0.0 to 0.043] | 0.012 [0.0 to 0.065]

33. Secondary Outcome: Culture-confirmed Invasive Disease (ID) Person Year Rate - In Children Starting Vaccination Within 7 Months of Life and Assigned to a 2-dose Primary Vaccination Course Till End of LT FU Period
Description: as for outcome 32
Time Frame: as for outcome 32
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Participants per 1000 person-years
Arm/Group | 10Pn2+1-6W-6M/043+053 Group | Ctrl-6W-6M/043+053 Group
Number analyzed (Participants) | 10053 | 10201
Participants per 1000 person-years
  Culture confirmed ID | 0.047 [0.013 to 0.122] | 0.268 [0.170 to 0.402]
  Pneumococcal invasive disease (IPD) | 0.024 [0.003 to 0.086] | 0.21 [0.124 to 0.331]
  Vaccine serotypes (vaccine type-IPD) | 0.012 [0.00 to 0.066] | 0.140 [0.072 to 0.244]
  Serotype 4 | 0.0 [0.0 to 0.044] | 0.0 [0.0 to 0.043]
  Serotype 6B | 0.0 [0.0 to 0.044] | 0.058 [0.019 to 0.136]
  Serotype 7F | 0.012 [0.0 to 0.066] | 0.0 [0.0 to 0.043]
  Serotype 14 | 0.0 [0.0 to 0.044] | 0.047 [0.013 to 0.119]
  Serotype 18C | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]
  Serotype 19F | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]
  Serotype 23F | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]
  Cross-reactive serotypes | 0.0 [0.0 to 0.044] | 0.047 [0.013 to 0.119]
  Serotype 6A | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]
  Serotype 19A | 0.0 [0.0 to 0.044] | 0.035 [0.007 to 0.102]
  Other pneumococcal serotypes | 0.012 [0.0 to 0.066] | 0.023 [0.003 to 0.084]
  Serotype 3 | 0.012 [0.0 to 0.066] | 0.012 [0.0 to 0.065]
  Serotype 12F | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]
  Serotype 15C | 0.0 [0.0 to 0.044] | 0.0 [0.0 to 0.043]
  H. influenzae ID | 0.012 [0.0 to 0.066] | 0.012 [0.0 to 0.065]
  Non-typeable (NTHI) | 0.012 [0.0 to 0.066] | 0.012 [0.0 to 0.065]
  Other bacteria | 0.012 [0.0 to 0.066] | 0.058 [0.019 to 0.136]
  Neisseria meningitidis | 0.012 [0.0 to 0.066] | 0.023 [0.003 to 0.084]
  Streptococcus pyogenes | 0.0 [0.0 to 0.044] | 0.023 [0.003 to 0.084]
  Moraxella catarrhalis | 0.0 [0.0 to 0.044] | 0.012 [0.0 to 0.065]

ADVERSE EVENTS:
Time Frame: SAEs were reported from Month 0 to end of blinded invasive disease (ID) phase (at least 30 months from study start), in 10PN-PD-DIT-043 subjects.
Description: Solicited and unsolicited AEs were not collected in this study.
Arm/Group | 10Pn3+1-6W-6M/043 Group | 10Pn2+1-6W-6M/043 Group | Ctrl-6W-6M/043 Group | 10Pn7-11M/043 Group | Ctrl7-11M/043 Group | 10Pn12-18M/043 Group | Ctrl12-18M/043 Group
All-Cause Mortality (participants affected / at risk) | 4/8427 | 4/9112 | 3/8872 | 0/3689 | 0/1812 | 0/6249 | 1/3020
Serious Adverse Events (participants affected / at risk) | 6/8427 | 7/9112 | 8/8872 | 3/3689 | 2/1812 | 2/6249 | 2/3020
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10Pn3+1-6W-6M/043 Group (N=8427) | 10Pn2+1-6W-6M/043 Group (N=9112) | Ctrl-6W-6M/043 Group (N=8872) | 10Pn7-11M/043 Group (N=3689) | Ctrl7-11M/043 Group (N=1812) | 10Pn12-18M/043 Group (N=6249) | Ctrl12-18M/043 Group (N=3020)
Kawasaki's disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gaucher's disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Krabbe's disease (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotonic-hyporesponsive episode (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden infant death syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reye's syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.